CLINICAL TRIAL: NCT03756064
Title: Neoadjuvant Study of Pyrotinib in Combination With Trastuzumab Plus Docetaxel and Carboplatin in Patients With HER2 Positive Early Stage or Locally Advanced Breast Cancer: a Single-arm, Ahead, Open-label Study
Brief Title: Neoadjuvant Study of Pyrotinib in Patients With HER2 Positive Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TCHP
Record Dates: First submitted 2018-11-21; First posted 2018-11-28 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Breast Cancer; Neoplasm, Breast; Breast Diseases
MeSH Terms: conditions — Breast Neoplasms; Breast Diseases | interventions — pyrotinib; Trastuzumab; Docetaxel; Carboplatin

STUDY DESIGN:
Intervention Model Description: Experimental: Pyrotinib (400mg orally daily)+Trastuzumab (8mg/kg iv load followed by 6mg/kg iv 3-weekly)+Docetaxel (75mg/m2)+ Carboplatin(AUC=5), for a total of 6 cycles.
  Placebo Comparator: Placebo Oral Tablet (400mg orally daily)+Trastuzumab (8mg/kg iv load followed by 6mg/kg iv 3-weekly)+Docetaxel (75mg/m2)+ Carboplatin(AUC=5), for a total of 6 cycles.
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Pyrotinib+Trastuzumab+Docetaxel +Carboplatin
  Interventions: Drug: Pyrotinib; Drug: Trastuzumab; Drug: Docetaxel; Drug: Carboplatin
- Control group (Placebo Comparator): Placebo Oral Tablet+Trastuzumab+Docetaxel +Carboplatin
  Interventions: Drug: Trastuzumab; Drug: Docetaxel; Drug: Carboplatin; Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Pyrotinib — Pyrotinib: 400mg orally daily
  Arms: Experimental group
Drug: Trastuzumab — Trastuzumab:8mg/kg iv load followed by 6mg/kg iv 3-weekly for a total of 6 cycles;
Drug: Docetaxel — Docetaxel: 75mg/m2 for a total of 6 cycles
Drug: Carboplatin — Carboplatin: AUC=5 for a total of 6 cycles
Drug: Placebo Oral Tablet — Placebo Oral Tablet: 400mg orally daily
  Arms: Control group

SUMMARY:
This is a randomized, double-blind multicenter Phase III study for evaluating the efficacy and safety of neoadjuvant pyrotinib and trastuzumab plus docetaxel and Carboplatin versus placebo and trastuzumab plus docetaxel and Carboplatin given as neoadjuvant treatment in HER2 positive early stage or locally advanced breast cancer.

DETAILED DESCRIPTION:
The investigators hypothesized that the experimental group (Pyrotinib+Trastuzumab+Docetaxel+ Carboplatin) could have a higher Pathological Complete Response (pCR) rate than the control group (Placebo +Trastuzumab+Docetaxel+ Carboplatin) in neoadjuvant chemotherapy.

It is proposed that 100 participants will be enrolled in this study. The target population is women with early breast cancer (stage of T1-4N0-3M0) who are eligible for primary systemic therapy.

The primary objective of the trial is to determine the pCR rate. The secondary objective of the trial is to determine the Event-free survival(EFS), Disease-free Survival (DFS), Distance Disease-free Survival (DDFS), Objective Response Rate (ORR) rate.

ELIGIBILITY:
Inclusion Criteria:

1. female patients, 18 years ≤ age ≤ 80 years；
2. Performance Status- Eastern Cooperative Oncology Group (ECOG) 0-1
3. Histologically confirmed invasive breast cancer（early stage or locally advanced）
4. HER2 positive (HER2+++ by IHC or FISH+)
5. Known hormone receptor status.
6. Cardiovascular: Baseline left ventricular ejection fraction (LVEF)≥55% measured by ECHO
7. Signed informed consent form (ICF)

Exclusion Criteria:

1. Metastatic disease (Stage IV) or inflammatory breast cancer
2. Previous or current history of malignant neoplasms, except for curatively treated: Basal and squamous cell carcinoma of the skin, Carcinoma in situ of the cervix.
3. Clinically relevant cardiovascular disease: Known history of uncontrolled or symptomatic angina, clinically significant arrhythmias, congestive heart failure, transmural myocardial infarction, uncontrolled hypertension ≥180/110);
4. Unable or unwilling to swallow tablets.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
pCR | through study completion, an average of 1 year
  Percentage of Participants With Pathological Complete Response (pCR) at the Time of Surgery.

SECONDARY OUTCOMES:
EFS | Following surgery until Year 3
  Event-free survival
DFS | Following surgery until Year 3
  Disease-free Survival
DDFS | Following surgery until Year 3
  Distance Disease-free Survival
ORR | Baseline up to cycle 4 (assessed at Baseline, at the time of pre-surgery)up to approximately 12 months
  Objective Response Rate

CONTACTS AND LOCATIONS:
Overall Officials: Ding Xiaowen, DR., Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ding Y, Mo W, Xie X, Wang O, He X, Zhao S, Gu X, Liang C, Qin C, Ding K, Yang H, Ding X. Neoadjuvant Pyrotinib plus Trastuzumab, Docetaxel, and Carboplatin in Early or Locally Advanced Human Epidermal Receptor 2-Positive Breast Cancer in China: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase 2 Trial. Oncol Res Treat. 2023;46(7-8):303-311. doi: 10.1159/000531492. Epub 2023 Jun 9. PMID 37302393